CLINICAL TRIAL: NCT00380809
Title: Rotational Atherectomy Prior to Taxus Stent Treatment for Complex Native Coronary Artery Disease. A Multicenter, Prospective, Randomized Controlled Trial.
Brief Title: Rotational Atherectomy Prior to Taxus Stent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Segeberger Kliniken GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SK 106
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Complex Calcified Coronary Lesions
MeSH Terms: interventions — Atherectomy, Coronary

ARMS (2):
- Rotational Atherectomy + PES (Active Comparator): Elective lesion preparation with rotational atherectomy priot to stent implantation
  Interventions: Procedure: Rotational Atherectomy + PES
- Standard Treatment (PES without Rotational Atherectomy) (Active Comparator): Stenting without prior rotational atherectomy, usually preceeded with balloon dilatation
  Interventions: Procedure: Standard Treatment (PES without Rotational Atherectomy)

INTERVENTIONS:
Procedure: Rotational Atherectomy + PES
  Arms: Rotational Atherectomy + PES
Procedure: Standard Treatment (PES without Rotational Atherectomy)
  Arms: Standard Treatment (PES without Rotational Atherectomy)

SUMMARY:
The primary purpose of this study is to evaluate the long term effects of the polymer-based slow-release paclitaxel-eluting stent (TAXUS; Boston Scientific), with or without prior rotablation, in an angiographically well defined group of patients with complex calcified coronary lesions.

DETAILED DESCRIPTION:
Calcification is an essential part of all atherosclerotic plaques. Its extent increases with the progression of atherosclerotic disease. Heavily calcified lesions form a particular threat to DES; both damage to the polymer coating during vigorous advancement and inadequate diffusion of the drug to the subintima through extensive calcium arcs could contribute to the ineffectiveness of DES when implanted into such lesions, or may lead to primary stent delivery or expansion failure. Rotational atherectomy can effectively ablate calcified plaques. In the DES era, data concerning rotational atherectomy are scarce. DES implantation following rotablation seems a rational combination, but is only poorly supported by controlled studies. In the present study, we are using the polymer-based slow-release paclitaxel-eluting stent (TAXUS; Boston Scientific), with or without prior rotablation, in an angiographically well defined group of patients with complex calcified coronary lesions. This prospective, randomized, controlled study aims at evaluating the long term effects of both strategies in this complex cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically proven coronary artery disease
* Angina II-IV° following the Canadian Cardiovascular Society Classification criteria and/or reproducible ischemia in the target area by ECG or scintigraphy
* The patient signing an informed written consent

From the following angiographic criteria, lesions must fulfil all first degree criteria and at least one second-degree criterion to be eligible for inclusion.

First degree criteria

* De-novo lesion in a native coronary artery
* Target reference vessel diameter between 2.5 and 4.0 mm by visual estimation
* Luminal diameter reduction of 70-99% by visual estimation
* Moderate to severe calcification of the target lesion (clearly defined)

Second degree criteria

* Ostial location
* Bifurcational lesions
* Long lesions (≥ 15mm)

Exclusion Criteria:

* Myocardial infarction within 4 weeks
* Left ventricular ejection fraction < 30%
* Limited long term prognosis due to other conditions

Angiographic exclusion criteria:

* Unprotected left main lesions
* Coronary artery bypass graft stenoses
* In-stent restenoses
* Chronic total occlusions
* Target vessel thrombus
* Target vessel dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss | 9 months

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | 9 months
In-segment late lumen loss | 9 months
In-segment binary restenosis | 9 months
Primary angiographic success | Immediate
Procedural duration and contrast dye amount | Immediate
Strategy success | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Gert Richardt, MD, Study Chair — Herz-Kreislauf-Zentrum Segeberger Kliniken GmbH; Ahmed A. Khattab, MD, Principal Investigator — Herz-Kreislauf-Zentrum Segeberger Kliniken GmbH; Mohamed Abdel-Wahab, MD, Principal Investigator — Herz-Kreislauf-Zentrum Segeberger Kliniken GmbH
Locations (1):
- Herz-Kreislauf-Zentrum Segeberger Kliniken GmbH, Bad Segeberg, Germany

REFERENCES:
- [Background] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. A polymer-based, paclitaxel-eluting stent in patients with coronary artery disease. N Engl J Med. 2004 Jan 15;350(3):221-31. doi: 10.1056/NEJMoa032441. PMID 14724301
- [Background] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. One-year clinical results with the slow-release, polymer-based, paclitaxel-eluting TAXUS stent: the TAXUS-IV trial. Circulation. 2004 Apr 27;109(16):1942-7. doi: 10.1161/01.CIR.0000127110.49192.72. Epub 2004 Apr 12. PMID 15078803
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Schofer J, Schluter M, Gershlick AH, Wijns W, Garcia E, Schampaert E, Breithardt G; E-SIRIUS Investigators. Sirolimus-eluting stents for treatment of patients with long atherosclerotic lesions in small coronary arteries: double-blind, randomised controlled trial (E-SIRIUS). Lancet. 2003 Oct 4;362(9390):1093-9. doi: 10.1016/S0140-6736(03)14462-5. PMID 14550694
- [Background] Warth DC, Leon MB, O'Neill W, Zacca N, Polissar NL, Buchbinder M. Rotational atherectomy multicenter registry: acute results, complications and 6-month angiographic follow-up in 709 patients. J Am Coll Cardiol. 1994 Sep;24(3):641-8. doi: 10.1016/0735-1097(94)90009-4. PMID 8077533
- [Background] Moussa I, Di Mario C, Moses J, Reimers B, Di Francesco L, Martini G, Tobis J, Colombo A. Coronary stenting after rotational atherectomy in calcified and complex lesions. Angiographic and clinical follow-up results. Circulation. 1997 Jul 1;96(1):128-36. doi: 10.1161/01.cir.96.1.128. PMID 9236427
- [Derived] Abdel-Wahab M, Richardt G, Joachim Buttner H, Toelg R, Geist V, Meinertz T, Schofer J, King L, Neumann FJ, Khattab AA. High-speed rotational atherectomy before paclitaxel-eluting stent implantation in complex calcified coronary lesions: the randomized ROTAXUS (Rotational Atherectomy Prior to Taxus Stent Treatment for Complex Native Coronary Artery Disease) trial. JACC Cardiovasc Interv. 2013 Jan;6(1):10-9. doi: 10.1016/j.jcin.2012.07.017. Epub 2012 Dec 19. PMID 23266232